CLINICAL TRIAL: NCT04803929
Title: Clinical Study of Autologous T Cells Modified With ILT3 Chimeric Antigen Receptor for Relapsed/Refractory Acute Myeloid Leukemia (M4/M5)
Brief Title: Clinical Study of Anti-ILT3 CAR-T Therapy for R/R AML(M4/M5)
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Carbiogene Therapeutics Co. Ltd. (Industry)
Collaborators: Zhejiang Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021KY014
Record Dates: First submitted 2021-03-15; First posted 2021-03-18 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: AML M4; AML M5
MeSH Terms: conditions — Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-ILT3 CAR-T cells (Experimental): All subjects were intravenous administrated with anti-ILT3 CAR-T cells
  Interventions: Biological: anti-ILT3 CAR-T

INTERVENTIONS:
Biological: anti-ILT3 CAR-T — Autologous T cells genetically modified with anti-ILT3 CAR

SUMMARY:
This study evaluates the safety and efficacy of novel ILT3-targeted CAR-T cell therapy for patients with relapsed or refractory acute myeloid leukemia (M4/M5).

DETAILED DESCRIPTION:
Our group has developed a novel anti-ILT3 CAR T cell therapy, and this pilot study is focused on the safety and efficacy of the anti-ILT3 CAR-T for R/R AML(M4/M5) patients. A total of 25 subjects are intravenously adminstered with anti-ILT3 CAR-T cells. The dosages of CAR-T cells follow the "3+3" dose increment program.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, aged ≥18 years or ≤70 years;
2. Acute myeloid leukemia AML M4/M5 subtype was diagnosed according to Fab standard classification, confirmed by bone marrow IHC or ILT3-positive expression by flow cytometry in monocytes (primary and young monocytes in bone marrow ≥20%)
3. Relapsed/refractory patients, whose conditions meet:

   * Recurrent AML diagnosis standard: complete remission (CR) after the original cells in peripheral blood again leukemia cells or bone marrow > 0.050 (with the exception of consolidation chemotherapy after bone marrow regeneration for other reasons) or myeloid leukemia cells infiltrating outside.
   * Refractory AML diagnostic criteria: after two standard regimen for treatment invalid early cure; patients who relapsed within 12 months after consolidation and intensive treatment after CR; relapsed after 12 months but failed to respond to conventional chemotherapy; 2 or more recurrences; patients with persistent extramedullary leukemia.
4. Main organ functions meet the following conditions:

   * Kidney function: creatinine clearance (absolute value) or 60 ml/min or creatinine < 2.0 mg/dl or < 2 times the subjects' age group upper limit of normal (ULN) blood.
   * Liver function: ALT ≤ 3 or less ULN, AST ≤ 3 or less ULN.
   * Heart function: the ejection fraction ≥ 50%, measured by echocardiography (ECHO) or more acquisition scan (MUGA).
   * Lung function: no clinical significance of pleural effusion, baseline blood oxygen saturation > 92%.
5. ECOG physical status score 0-3.
6. No use of steroid hormones within 2 weeks.
7. Sufficient venous access to single or venous blood collection is available, and there are no other contraindications to blood cell separation.
8. Signed written informed consent form.

Exclusion Criteria:

Subjects will not be included in the study if they meet any of the following criteria:

1. Pregnant or lactating women;
2. HIV serological positive;
3. Active bacterial, fungal or viral infections that are not controlled by treatment;
4. Suffer from coronary heart disease, angina pectoris, myocardial infarction, arrhythmia, cerebral thrombosis, cerebral hemorrhage or other serious cardiovascular and cerebrovascular diseases;
5. History and concomitant diseases:

   * Subjects with known or suspected autoimmune diseases or immunodeficiency diseases;
   * Subjects requiring systemic treatment with corticosteroids or other immunosuppressive agents during treatment;
   * Subjects who have previously received other gene therapies;
   * Subjects with a history of organ transplantation (referring to solid organ transplantation);
   * Subjects with severe mental disorders;
   * Participated in other clinical studies within one month before the collection of PBMC;
   * Uncontrolled active hepatitis B and/or C infection (hepatitis B: HBV DNA > 500 IU/ml or copy number > 2500 copies /ml;
   * Hepatitis C: HCV antibody positive and HCV-RNA levels above the detection limit);
   * Any serious or uncontrolled disease that the Investigator considers to be likely to increase the risk associated with study participation, study drug administration, or affect the subject's ability to receive the study drug;
   * Subjects who underwent major surgery or suffered significant trauma within 4 weeks prior to the collection of PBMCs, or who are expected to require major surgery during the study period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-03-03 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Rate of grade 3 or 4 treatment related adverse effects | up to 24 weeks after first infusion
  All the CAR-T treatment related adverse events，including Dose limiting toxicity (DLT), cytokine release syndrome (CRS), CAR-T associated encephalopathy syndrome, will be assessed and graded by NCI CTCAE v 5.0.
Implantation endpoint | up to 2 years after first infusion
  To assess the duration of CAR-positive T cells in circulation, the copy number of CAR DNA was measured at the preset follow-up time point. The time when the results of any two consecutive tests were negative, were recorded as the "implantation endpoint"

SECONDARY OUTCOMES:
Disease specific response | up to 2 years after first infusion
  Disease specific response includes, but are not limited to, complete response (CR) including morphological leukemia-free status, morphological CR, cytogenetic CR, molecular CR, and partial response (PR).
Overall survival | up to 2 years after inclusion
  From date of inclusion to date of progression, relapse, or death from any cause
Progress-free survival | up to 2 years after inclusion
  The length of time that a participant's disease did not progress during and after CAR-T treatment
CAR-T residue | up to 2 years after first infusion
  The residue of CAR-positive T cells in circulation determined by flow cytometry
Minimal residual disease (MRD) | up to 2 years after first infusion
  MRD is a status that none tumor cells can be detected by standard cell morphology.

CONTACTS AND LOCATIONS:
Overall Officials: Jianping Lan, Principal Investigator — Zhejiang Provincial People's Hospital
Locations (1):
- Zhejiang Provincal People's Hospital, Hangzhou, Zhejiang, China